CLINICAL TRIAL: NCT05429931
Title: Urdu Version of The Ronald Morris Disability Questionnaire in Patients With Low Back Pain : Assessing Its Psychometric Properties and Cultural Adaptation.
Brief Title: Reliability and Validity of Urdu Version of Ronald Morris Disability Questionnaire in Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0296
Record Dates: First submitted 2022-06-20; First posted 2022-06-23 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: Ronald Morris Disability Questionnaire; Urdu Version; Reliability; Validity; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose of this Research is to convert Ronald Morris Disability Questionnaire into Urdu language and check the accuracy and logic in Pakistani low back pain population. Also check its correlation with Oswestry Disability Index and Visual Analogue Scale.

DETAILED DESCRIPTION:
The Ronald Morris Disability Questionnaire will be translated into Urdu and culturally adapted for people with low back pain. Ronald Morris Disability Questionnaire will be given to 80 people who will be chosen by using a convenient sampling method. Method of sampling based on pre-determined inclusion and exclusion criteria. To examine intra-observer reliability of the final Ronald Morris Disability Questionnaire, two observers will fill out Oswestry Disability Index and Visual Analogue Scale questionnaires on the same day to test inter-observer evaluation. After 30 minutes of the initial treatment, the second application will be applied. The first observer will do the third assessment after seven days. Statistical Package of Social Sciences Version 24 will be used to enter and analyse data. The alpha value of Cronbach's alpha will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Average Age of patient 48 years.
* Patient with chronic low back pain have at least 3 month duration .
* Patient with mechanical Low Back Pain

Exclusion Criteria:

* Patient with non - mechanical Low Back Pain
* Patient have neurological deficits .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pakistani population with Chronic Low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Disability Questionnaire | 1st day
  Roland-Morris Disability Questionnaire consist of 24 point according to low back pain population in which patients tell about all Daily Activity . patients scores the questionnaire among 24 points. Roland-Morris Disability Questionnaire is the highest result possible '24'.
Oswestry Disability Index | 1st day
  Oswestry Disability Index is an instrument or scale use for the evaluation of pain . this scale is especially designed for low back pain.
  Oswestry Disability Index consist of 10 section or 9 section divide the point out of 50 or 45 . if one section is not score then divided by 45 and get score of patient.after get score multiply with 100 to get percentage. 0 to 21% indicate minimal disability , 21 to 40 indicate moderate disability and 41 to 60 indicate severe disability. 61 to 80 indicate crippled.
Visual Analogue Scale | 1st day
  Visual analog scale is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No